CLINICAL TRIAL: NCT06193681
Title: The Efficiency of Supervised Exercise Program Versus Personalized Mobile-Based Exercise Program in Patients With Juvenile Idiopathic Arthritis
Brief Title: Efficiency of Supervised Exercise Program Versus Mobile-Based Exercise Program in Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Asena Yekdaneh, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAYekdaneh1
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Adolescents; Juvenile Idiopathic Arthritis; mobile application; ehealth; exercise; personalized exercise; mhealth
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pedi@ctivity Exercise Mobile Application (Experimental)
  Interventions: Other: Pedi@ctivity Exercise Mobile Application Exercise Program
- Supervised Exercise Group (Experimental)
  Interventions: Other: Supervised Exercise Group

INTERVENTIONS:
Other: Pedi@ctivity Exercise Mobile Application Exercise Program — The first group of the study received a mobile application (Pedi@ctivity) based exercise program. With the Pedi@ctivity exercise mobile application, the selected exercises and exercise program will be offered personalized to each adolescent for 12 weeks. After 12 weeks, the effectiveness of the Pedi@ctivity mobile application-based exercise program on the evaluation parameters will be investigated.
  Arms: Pedi@ctivity Exercise Mobile Application
Other: Supervised Exercise Group — In the physiotherapist-supervised personalized exercise program, the exercises selected through the Pedi@ctivity exercise mobile application will be applied to adolescents under the supervision of a physiotherapist (2 sessions face-to-face, 1 session online/synchronous).
  Arms: Supervised Exercise Group

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is a heterogeneous, idiopathic, chronic inflammatory, rheumatic disease that is most common in childhood and is thought to involve immunological mechanisms in its etiopathogenesis. Exercise and physical activity (PA) approaches have an important place in the treatment of childhood rheumatic diseases. These approaches alleviate both the symptoms of children and adolescents' chronic diseases and complications secondary to pharmacological treatments, and prevent the occurrence of new chronic diseases. However, it is difficult to draw conclusions regarding the effects of exercise types on patients with JIA, as there are few comparative studies in the literature investigating the superior effects of exercise programs on disease-specific problems.

Physical, individual, social and psychological factors that create barriers to PA and exercise participation in children and adolescents with rheumatic disease significantly affect PA and exercise adherence. In this regard, online applications stand out as an important strategy for encouraging behavioral change, providing motivational and social support, and allowing feedback and interaction with health professionals using information and communication technologies.

It is emphasized that digital health applications should be designed more comprehensively and personalized to increase participation in PA promotion and regular exercise programs and be compared with control group exercise programs in order to increase their usability in this disease population and examine their effectiveness.

This study will be planned as a randomized controlled study. Adolescent JIA patients between the ages of 12-18 will be included in the study and will be divided into 2 groups. The first group will receive a personalized exercise program under the supervision of a physiotherapist, 3 sessions per week (2 session face to face, 1 session online) for 12 weeks. A personalized mobile application-based exercise program will be applied to the second group for the same week and frequency. This study can contribute to the literature by investigating effective methods in improving physical fitness, physical activity, walking and balance functions in patients with JIA.

Adolescents in both groups will be given smart watches to promote PA and monitor health parameters. The evaluation periods for both groups are stated below; T0: Start T1: Before the exercise program (after 3 months of PA monitoring with a smart watch) T2: It will be carried out after the exercise program (12 weeks later). The effectiveness of the exercise program to be applied on the evaluation parameters will be demonstrated by comparing the two groups after the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Being 12-18 years old
* Being diagnosed with JIA at least 6 months ago at the Istanbul Medical Faculty Pediatric Rheumatology Clinic
* Being diagnosed with Oligoarticular/Polyarticular JIA
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of trauma or surgery affecting the musculoskeletal system in the last 6 months
* Having an additional chronic disease affecting the musculoskeletal system
* Having vision or hearing problems
* Having a level of cognitive impairment that cannot understand the commands given

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
FitnessGram Physical Activity Test Battery-Progressive Aerobic Cardiovascular Endurance Running (PACER) | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  PACER is an adapted version of the 20 meter shuttle run test and is a field test consisting of multiple stages. The participant will run back and forth in a 20 meter area accompanied by the music coming from the voice recorder. The beep indicates when the participant should finish a lap. The test will start at slow speeds and will gradually increase each minute. The test will be terminated when the participant cannot continue to run at the level he has reached. The number of laps completed at the end of the test will be recorded. PACER is a more fun alternative to other distance running tests. It is recommended for use in children, adolescents and young adults. PACER will be used to assess the aerobic capacity of adolescents.
FitnessGram Physical Activity Test Battery-Curl-up Test | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  The participant will begin the test in the supine position, knees flexed approximately 140 degrees, feet flat on the floor, and legs slightly apart. The participant's arms will be parallel to the floor and torso. The palm will be positioned on the floor with the fingers stretched out. The purpose of this test is to do as many sit-ups as possible at a given speed. A maximum of 75 shuttles counts. The number of shuttles performed at the end of the test will be recorded. The curl-up test will be used to evaluate the abdominal muscle strength and endurance of adolescents.
FitnessGram Physical Activity Test Battery-Trunk Lift Test | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  The participant will begin the test in the prone position with their hands placed under the thigh. A sign will be placed on the floor at the participant's eye level. During the movement, the participant will focus on this sign. During the test, the participant slowly and in a controlled manner raises their torso to a maximum height of 12 inches. The head is kept in neutral alignment with the spine. At the end of the test, the distance between the floor and the participant's chin will be measured with a ruler and the score will be recorded in centimeters (cm). Trunk lift test will be used to evaluate trunk extensor muscle strength and flexibility of adolescents.
FitnessGram Physical Activity Test Battery-Push-up Test | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  The participant will begin the test in the prone position, with their hands shoulder-width or wider than shoulder-width apart, fingers stretched, palms on the floor, and legs slightly apart. During the test, the participant lowers his torso towards the ground and raises himself up again when his elbows are bent 90º. The movement is repeated as much as possible. The rhythm is set to 20 push-ups per minute or 1 push-up per 3 seconds. The test is terminated when the participant makes a mistake twice. The number of push-ups performed at the end of the test will be recorded. The push-up test will be used to evaluate the upper extremity muscle strength and endurance of adolescents.
FitnessGram Physical Activity Test Battery-Back Saver Sit and Reach Test | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  During the test, the participant takes off his shoes and sits in front of the test apparatus. A box is needed for the test. This box is 35 cm long, 45 cm wide, 32 cm high. A top plate 55 cm long and 45 cm wide is put on top of the box. One leg of the participant is completely straight while the other is bent at the knee. The participant reaches forward four times with their hands on top of each other, holding the fourth reach position for 1 second. At the end of the test, the distance traveled will be recorded. The Back Saver Sit and Reach Test will be used to evaluate the hamstring flexibility of adolescents.
6 Minute Walk Test (6 MWT) | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  The 6-minute walk test is a well-tolerated, easy-to-apply and simple test that shows the submaximal level of functional capacity. This test measures the distance that participants can walk quickly on a hard and flat surface in 6 minutes. Participants rest in a chair near the starting position for at least 10 minutes before the start of the test. Before and after the test, heart rate, blood pressure, saturation are measured, and fatigue level is determined with the Modified Borg scale. Participants are told how to perform the test. At the end of the test, the distance walked by the participants in 6 minutes will be recorded in meters. The 6 Minute Walk Test will be used to evaluate the functional capacities of adolescents.
10 Stairs Climbing Test | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  During the test, participants will be asked to climb 10 steps (14x28x120cm) as fast as possible. Step climbing times will be measured in seconds with a stopwatch. The 10 Step Climbing Test will be used to evaluate the functional capacity of adolescents.
1 Minute Sit to Stand Test | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  We will ask the patient to sit in a chair where she/he can stand upright, and then, with the help of a stopwatch, we will record the number of times she/he sits down and stands up from the chair in 1 minute.

SECONDARY OUTCOMES:
Heart Rate | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  Heart rate includes in the health parameters. The adolescents included in the study will be given a smart watch and will be asked to use the watches for 3 months to record. With wearable activity tracker watches, data on the person's heart rate (beats per minute) during the day will be recorded.
Number of steps | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  Number of steps includes in the health parameters. The adolescents included in the study will be given a smart watch and will be asked to use the watches for 3 months. With wearable activity tracker watches, data on the number of steps taken per day (step count in numbers) will be recorded.
Oxygen saturation | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  Oxygen saturation includes in the health parameters. Oxygen saturation is a measure of how much hemoglobin is currently bound to oxygen compared to how much hemoglobin remains unbound. The adolescents included in the study will be given a smart watch and will be asked to use the watches for 3 months. With wearable activity tracker watches, data on the person's oxygen saturation (%) will be recorded.
Daily calories | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  Daily calories includes in the health parameters. The adolescents included in the study will be given a smart watch and will be asked to use the watches for 3 months. With wearable activity tracker watches, data on the daily calories burned (cal in numbers) will be recorded.
Activities | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  Daily activities includes in the health parameters. The adolescents included in the study will be given a smart watch and will be asked to use the watches for 3 months. With wearable activity tracker watches, data on the daily performed activities and locations will be recorded.
KFORCE Plates | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  KFORCE Plates is a force platform used to improve balance and evaluate lower extremity muscle symmetry and strength. It consists of two independent plates. KFORCE plates allow measurement of static and dynamic balance in a wide range of movements. It can also determine the center of gravity and measure weight distribution during the stance phase. It evaluates squatting, push-up and jumping characteristics and provides a report containing multiple data as a result of the measurement. Static and dynamic balance analyzes of adolescents will be performed with the device.
KFORCE Muscle Controller | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  KFORCE Muscle Controller is a hand dynamometer used to evaluate muscle strength. It evaluates maximum strength, endurance and muscle symmetry. The muscle controller is versatile and can be adapted to many configurations. As a result of the evaluation, the participant's results are recorded in a database. The participant's progress can then be followed in the application's database (13). The muscle strength of adolescents will be evaluated with the device.
Digitsole Pro® system | Change from Baseline, Before the exercise program (after 3 months of PA monitoring with a smart watch) and after the exercise program (12 weeks later).
  Digitsole Pro® system consists of wireless sensors, can be fitted in to any shoe and offer the ability to measure spatial, temporal, and kinematic gait parameters. The intelligent insoles feature several sensors that detect and capture foot movements and a micro process or that calculates gait related biomechanical data. Each PODOSmart®insole has an inertial platform that records each foot's walking steps, running strides, and orientations in space with sampling frequency of 208 Hz for walk analysis.The Bluetooth connection box retrieves the collected data by the smart insoles. Then, those data are processed by proprietary artificial intelligence algorithms to calculate the spatiotemporal, kinematic, and biomechanical parameters. Participants' features of walking will be evaluated with the Digitsole Pro® system.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Assoc. Prof., Study Chair — Istanbul University-Cerrahpaşa, Faculty of Health Science, Department of Physiotherapy and Rehabilitation; Nuray Aktay Ayaz, Prof. Dr., Study Chair — Istanbul Faculty of Medicine, Department of Internal Medicine, Department of Pediatric Rheumatology; Asena Yekdaneh, Principal Investigator — Istanbul University-Cerrahpasa, Institute of Postgraduate Education
Locations (1):
- Istanbul University-Cerrahpasa, Institute of Postgraduate Education, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No